CLINICAL TRIAL: NCT04301505
Title: Checklist Based Method for Improvement of COPD Care in Elderly in General Practice: Cluster Randomized Controlled Trial Using Electronic Health Records
Brief Title: Improvement in COPD Elderly Patients Health: Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016/21/B/NZ7/02052
Record Dates: First submitted 2020-02-18; First posted 2020-03-10 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease (COPD); elderly; exacerbation of COPD; prevalence; checklist; randomized controlled trial; electronic health records
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): Usual care.
- Intervention 1 (Other): COPD management checklist will be delivered at the beginning of the study.
  Interventions: Other: Intervention 1
- Intervention 2 (Other): COPD management checklist will be delivered at the beginning of the study and repeated after 6 months.
  Interventions: Other: Intervention 2

INTERVENTIONS:
Other: Intervention 1 — Checklist will be delivered at the beginning of the study. The educational intervention program will consist of a checklist that provides family physicians with COPD management for the elderly.
  Arms: Intervention 1
Other: Intervention 2 — The same checklist will be delivered at the beginning of the study and repeated after 6 months.
  Arms: Intervention 2

SUMMARY:
Guidelines development, their implementation and the physicians' adherence may have an impact on the occurrence of Chronic Obstructive Pulmonary Disease (COPD) exacerbations and patient's quality of life. We have developed an educational program based on a checklist to assist general practitioners in managing COPD patients. The results of this trial based on electronic health records from BIG DATA databases, such as the electronic health record (EHR) of patients from the National Health Found, associated with checklist, will be directly applicable to primary care in Poland and add new data to the growing body of evidence on interventions to improve chronic illness care and patient's quality of life.

DETAILED DESCRIPTION:
This study is the three-arm cluster controlled randomized trial (CRT) with the patients nested within practices. The effectiveness of Checklist in reduction of COPD exacerbations health outcomes in COPD patients after 2 interventions will be evaluated and compared to that of usual care. The results of this trial will be directly applicable to primary care in Poland and add new data to the growing body of evidence on interventions to improve chronic illness care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients: aged 65 years and older with diagnosis of COPD registered as J-44 (ICD-10).
2. Centres: Primary Health Care Centers (PHCC) with at least 46 COPD patients listed.

Exclusion Criteria:

None

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2520 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
The proportion of elderly patients hospitalized with the J-44 code as a main reason for admission after interventions vs. control. | 12 months
  Variables from BIG DATA databases, such as the electronic health record (EHR) of patients from the National Health Found, associated with checklist will be used to assess hospitalization of elderly patients with the J-44 code as a main reason for admission after 1 year.

SECONDARY OUTCOMES:
The proportion of deaths, or specific short and long acting drugs prescribed in intervention arms vs. control and the effect of the educational intervention. | 12 months
  Variables from BIG DATA databases, electronic health records (EHR) associated with checklist will be used to assess patients' health outcomes.
  The effect of the educational intervention will be evaluated using logistic 2-level regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Maciek Godycki-Cwirko, Prof., Principal Investigator — Centre for Family and Community Medicine, Medical Univeristy of Lodz, Poland
Locations (1):
- Medical University of Lodz, Lodz, Poland

REFERENCES:
- [Derived] Kowalczyk A, Zakowska I, Andrzejewska E, Kosiek K, Godycki-Cwirko M. A checklist-based method for improving COPD care for the elderly in general practice: study protocol for a cluster randomized controlled trial using electronic health records. Trials. 2021 Feb 25;22(1):161. doi: 10.1186/s13063-021-05103-0. PMID 33632282